CLINICAL TRIAL: NCT00768937
Title: Sorafenib as Inhibitor of Collateral Tumor Vessel Growth During Transarterial Chemoembolisation (TACE) for Hepatocellular Carcinoma (HCC)- a Pilot Trial to Evaluate Safety and Biological Response
Brief Title: Sorafenib and Transarterial Chemoembolization for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Univ. Prof. Dr. Markus Peck-Radosavljevic, Abteilung Gastroenterologie und Hepatologie, Medizinische Universität Wien
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SORATACE1
Record Dates: First submitted 2008-10-03; First posted 2008-10-08 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; sorafenib; transarterial chemoembolization; tumor angiogenesis; angiogenic factors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): all patients will be treated with sorafenib
  Interventions: Drug: Sorafenib; Procedure: Transarterial chemoembolisation (TACE)

INTERVENTIONS:
Drug: Sorafenib — All patients will receive Sorafenib (800 mg/day) p.o. beginning two weeks before the first TACE and every day thereafter until patient death or premature withdrawal from study.
  Other Names: Nexavar (brand name)
Procedure: Transarterial chemoembolisation (TACE) — TACE will be carried out with doxorubicin (75 - 50 - 25 mg/m2, depending on serum bilirubin levels ≤ 1.5, 1.5 - 3, 3 - 5 mg/dL) : lipiodol (1:1) in a total volume of 20 mL; after administration of doxorubicin:lipiodol, additional embolisation will be carried out with bead block-endospheres. TACE will be repeated every 4 weeks for 3 cycles; additional cycles will be offered if clinically indicated (but no PEI or RF-ablation should be carried out after inclusion into the study)

SUMMARY:
Hepatocellular carcinoma (HCC) as the third most common cause of cancer-related death has a very poor prognosis. Aim of this open label single arm non randomized pilot trial is the evaluation of the efficacy and safety of sorafenib in combination with TACE in patients with unresectable HCC. Efficacy ad safety will be compared with a historical TACE-only group of a placebo controlled TACE-trial.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) as the third most common cause of cancer-related death has a very poor prognosis.

Aim 1: Efficacy of Sorafenib in combination with TACE TACE is an established therapy for patients with unresectable HCC and has been shown to significantly improve survival in these patients compared to no treatment. Quite often after cutting off the blood supply through the hepatic artery, the tumor induces active angiogenesis to promote collateral blood vessel growth from liver capsule arteries or collaterals from the gastroduodenal artery leading to tumor recovery and proliferation. Inhibition of this neoangiogenetic and proliferation activity after TACE by the multikinase inhibitor Sorafenib, already approved for HCC, could lead to significantly improvement in tumor control and survival in patients with advanced stage HCC.Safety will be compared with a historical TACE-only group of a placebo controlled TACE-trial.

Aim 2: Safety of Sorafenib in combination with TACE:

So far there are no reports about the safety of Sorafenib in combination with TACE. Here we evaluate the safety and tolerability of this combination until 12 weeks after the last TACE.

Aim 3: PPG-Measurement:

Development of portal hypertension in cirrhosis occurs due to two main pathophysiologic mechanisms: the increase in resistance to portal blood flow resulting from increased intrahepatic resistance and the decreased arteriolar vascular tone in the splanchnic vascular bed leading to increased splanchnic inflow of blood. Very recently, it has been shown that increased splanchnic inflow does not only result from arteriolar vasodilation due to excess NO-production in the splanchnic vascular bed but also from an increase in neoangiogenesis in the splanchnic circulation. Increased neovessel formation occurred within a few days of onset of portal hypertension both in a cirrhotic and an extrahepatic murine model of portal hypertension. Neoangiogenesis was effectively inhibited by either an antibody against VEGF-R2 or an inhibitor of VEGF-R2 autophosphorylation, resulting in a reduction of splanchnic blood flow.

Most recently, a combination of a VEGF and a PDGF blocker further decreased portal pressure in an experimental preclinical model.

As Sorafenib is a VEGF and PDGF blocker, we aim to analyze the influence of Sorafenib on portal hypertension and systemic and hepatic hemodynamics.

Aim 4: Biomarkers for treatment response:

Furthermore, we aim to analyze methylated tumor DNA in serum of patients with HCC undergoing Sorafenib treatment and TACE as possible marker of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed HCC not suitable for OLT or resection ( > 3 nodules, >5 cm diameter, vascular invasion, clinically significant portal hypertension, other contraindications against OLT)
* Child-Pugh Stage A or B
* Liver disease of any etiology
* Written informed consent (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures
* Patient must be able to comply with the protocol
* Age ≥ 18 years
* Women of childbearing potential must have a negative serum pregnancy test done 1 week prior to the administration of the Sorafenib.

Fertile women and men of childbearing potential ( < 2 years after last menstruation in women) must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)

* Haematology:

Absolute neutrophil count (ANC) > 1 x 109/L Platelet count > 40 x 109/L Haemoglobin > 9 g/dL (may be transfused to maintain or exceed this level) Prothrombin time ≥ 40%

* Biochemistry:

Total bilirubin < 5 mg/dL Serum creatinine < 3.0 mg/dL

* Life expectancy of > 3 months

Exclusion Criteria:

* Extrahepatic tumor spread
* Complete portal vein thrombosis (common trunk)
* Child-Pugh-Stage C
* Prior TACE or TAE
* Other experimental therapies for HCC
* Acute variceal bleeding within the last 2 weeks
* Large oesophageal varices ( > 5 mm diameter) without prophylactic band ligation
* Past or current history (within the last 2 years prior to randomisation) of malignancies except for the indication under this study and curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., seizure not controlled with standard medical therapy or history of stroke within < 6 months), excluding hepatic encephalopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants for therapeutic purposes
* Chronic, daily treatment with aspirin (>325mg/day)
* Pregnancy (positive serum pregnancy test) or lactation
* Uncontrolled hypertension
* Serious, non-healing wound, ulcer, or bone fracture
* Currently or recent (within the 30 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents ( ≤ 6 months prior to study entry), myocardial infarction ( ≤ 6 months prior to study entry), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of Sorafenib/TACE or patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Time to Progression (Efficacy) | Until disease progression
Safety of Sorafenib in combination with TACE | Continuously until 12 weeks after the last TACE

CONTACTS AND LOCATIONS:
Overall Officials: Markus Peck-Radosavljevic, Prof. Dr., Principal Investigator — Abteilung Gastroenterologie und Hepatologie, Medizinische Universität und AKH Wien
Locations (1):
- Abteilung Gastroenterologie und Hepatologie, Medizinische Universität und AKH Wien, Vienna, Austria